CLINICAL TRIAL: NCT04211272
Title: A Single-center, Open-label, Single-sequence, 2-part Study to Investigate the Effect of 75 mg Macitentan Once Daily at Steady State on the Pharmacokinetics of Riociguat, Sildenafil, Rosuvastatin and Tadalafil in Healthy Male Subjects
Brief Title: A 2-part Study to Investigate the Effect of Macitentan in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CR108727; 2019-004001-27 (EudraCT Number); 67896062PAH1003 (Other: Actelion)
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — macitentan; Sildenafil Citrate; riociguat; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: Macitentan + Substrate Drug (Sildenafil/Riociguat) (Experimental): Participants will receive a single dose of film-coated tablet of sildenafil under fasted condition (Treatment A1), then riociguat under fasted condition (Treatment A2) followed by macitentan under fed condition (Treatment B1), then riociguat along with macitentan under fasted conditions followed by macitentan under fed conditions (Treatment B2) and then sildenafil along with macitentan under fasted condition (Treatment B3). Macitentan will be administered in an up-titration regimen.
  Interventions: Drug: Macitentan; Drug: Sildenafil; Drug: Riociguat
- Part B: Macitentan + Substrate Drug (Rosuvastatin) (Experimental): Participants will receive a single dose of film-coated tablet of rosuvastatin under fasted condition (Treatment A1), then macitentan under fed condition (Treatment B1) followed by rosuvastatin along with macitentan under fasted condition followed by macitentan under fed condition (Treatment B2). Macitentan will be administered in an up-titration regimen. Part B of the study will be conducted depending on the results of Part A and feedback from Health Authorities.
  Interventions: Drug: Macitentan; Drug: Rosuvastatin

INTERVENTIONS:
Drug: Macitentan — Macitentan will be administrated as film-coated tablet in Part A and Part B.
  Other Names: JNJ-67896062-AAA
Drug: Sildenafil — Sildenafil will be administrated as film-coated tablet in Part A.
  Other Names: Revatio
  Arms: Part A: Macitentan + Substrate Drug (Sildenafil/Riociguat)
Drug: Riociguat — Riociguat will be administrated as film-coated tablet in Part A.
  Other Names: Adempas
  Arms: Part A: Macitentan + Substrate Drug (Sildenafil/Riociguat)
Drug: Rosuvastatin — Rosuvastatin will be administrated as film-coated tablet in Part B.
  Other Names: Crestor
  Arms: Part B: Macitentan + Substrate Drug (Rosuvastatin)

SUMMARY:
The purpose of this study is to evaluate the effect of macitentan at steady state on the pharmacokinetic (PK) of a single dose of riociguat and sildenafil (Part A); and rosuvastatin (Part B) when co-administered to healthy male participants under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male (according to their reproductive organs and functions assigned by chromosomal complement)
* Healthy on the basis of physical examination, medical history, and 12 lead electrocardiogram (ECG) performed at screening. This determination must be recorded in the participant's source documents and initialed by the investigator
* Body mass index (BMI; weight per height^2) between 18.0 and 30.0 kilogram (kg)/meter square (m^2) (inclusive), and body weight not less than 50.0 kg at screening and on Day -5
* Blood pressure (after the participant is supine for 5 minutes) between 100 and 140 millimeters of mercury (mmHg) systolic blood pressure (SBP), inclusive, and between 60 and 90 mmHg Diastolic blood pressure (DBP), inclusive, at screening and on Day -5. If blood pressure is out of range, up to 2 repeated assessments are permitted
* Heart rate between 45 and 90 beats per minute (bpm, inclusive) at screening and on Day -5

Exclusion Criteria:

* History of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, which is considered cured with minimal risk of recurrence)
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for paracetamol (acetaminophen) within 14 days before the first dose of the study drug is scheduled until completion of the study
* A participant who has been on a known cytochrome P450 (CYP) inhibitor or inducer or transport inhibitor or inducer should be excluded from the study based upon the duration of the inhibitor or inductive effect and also at least 5 terminal half-lives of the drug, vitamin or herbal supplements
* Orthostatic hypotension (greater than [>] 20 mmHg decrease in SBP or >10 mmHg decrease in DBP after 2 minutes of standing compared to supine blood pressure)
* One or more of the following lab abnormalities at screening, defined as grade 1 or more by the World Health Organisation (WHO) Toxicity Grading Scale for Determining the Severity of Adverse Events, February 2003: aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than or equal to (>=) 1.25 * upper limit of normal (ULN), total bilirubin >=1.25 * ULN, and Hemoglobin less than or equal to (<=) 10.5 gram per deciliter (g/dL)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

PRIMARY OUTCOMES:
Part A and Part B: Area Under the Plasma Analyte Concentration-time Curve from Time Zero to Infinite Time (AUC[0-infinity]) of Sildenafil, Riociguat, Rosuvastatin | Up to 25 days
  AUC(0-infinity) is defined as area under the plasma analyte concentration-time curve from time 0 to infinite time.
Part A and Part B: Maximum Observed Plasma Analyte Concentration (Cmax) of Sildenafil, Riociguat, Rosuvastatin | Up to 25 days
  Cmax is defined as the maximum observed plasma analyte concentration.

SECONDARY OUTCOMES:
Part A: Area Under the Plasma Analyte Concentration-time Curve from Time Zero to Infinite Time (AUC[0-infinity]) of Desmethyl-sildenafil, M1 (Metabolite of Riociguat) and ACT-132577 (Metabolite of Macitentan) | Up to 25 days
  AUC(0-infinity) is defined as area under the plasma analyte concentration-time curve from time 0 to infinite time.
Part A: Maximum Observed Plasma Analyte Concentration (Cmax) of Desmethyl-sildenafil, M1 and ACT-132577 | Up to 25 days
  Cmax is defined as the maximum observed plasma analyte concentration.
Part A and Part B: Area Under the Plasma Analyte Concentration-time Curve from 0 to Time t of the Last Measured Concentration (AUC[0-t]) of Sildenafil, Desmethyl-sildenafil, Riociguat, M1, Macitentan, ACT-132577, Rosuvastatin | Up to 25 days
  AUC(0-t) is defined as area under the plasma analyte concentration-time curve from time 0 to time t of the last measured concentration above the lower limit of quantification (LLOQ), calculated according to the linear trapezoidal rule, using the measured concentration-time values above the LLOQ.
Part A and Part B: Time to Reach Maximum Observed Plasma Analyte Concentration (Tmax) of Sildenafil, Desmethyl-sildenafil, Riociguat, M1, Macitentan, ACT-132577, Rosuvastatin | Up to 25 days
  Tmax is defined as actual sampling time to reach maximum observed plasma analyte concentration.
Part A and Part B: Apparent Elimination Half-life (t1/2) of Sildenafil, Desmethyl-sildenafil, Riociguat, M1, Macitentan, ACT-132577, Rosuvastatin | Up to 25 days
  t1/2 is defined as the time measured for the plasma concentration to decrease by 1 half of its original concentration. It is associated with the terminal slope of the semilogarithmic drug concentration-time curve, calculated as t1/2=0.693/ lambda(z).
Part A and Part B: Trough Plasma Concentration (Ctrough) of Macitentan and ACT-132577 | Up to 25 days
  Ctrough is defined as the observed plasma concentration before dosing or at the end of the dosing interval.
Part B: Number of Participants with Adverse Event as a Measure of Safety and Tolerability | Up to Day 45
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Actelion Clinical Trial, Study Director — Actelion
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency